CLINICAL TRIAL: NCT04801212
Title: The Effects of Lumbar Stabilization Exercises With and Without Jaw Movements in Non-specific Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Khan, Principal Investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2021-02-03; First posted 2021-03-16 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Chronic Nonspecific Low Back Pain; Core Stability; Jaw Movements; Temporomandibular Joint

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stability exercises with teeth clenching (Experimental): The intervention frequency will be 2 sessions per week for the duration of 6 weeks, comprising of 45 minutes session. Both groups will receive heat pack on lumbar spine for 12 minutes and both interventions will be held under the supervision of qualified Musculoskeletal Physiotherapists. During intervention and after 6 weeks of intervention, both groups will be given a home exercise program consist of same exercises they have carried out in the clinic for the duration another 6 weeks. The participants will be asked to keep diaries of their exercises they have carried out each week.
  Interventions: Other: core stability exercises with teeth clenching; Other: core stability exercises
- core stability exercises alone (Active Comparator): The intervention frequency will be 2 sessions per week for the duration of 6 weeks, comprising of 45 minutes session. Both groups will receive heat pack on lumbar spine for 12 minutes and both interventions will be held under the supervision of qualified Musculoskeletal Physiotherapists. During intervention and after 6 weeks of intervention, both groups will be given a home exercise program consist of same exercises they have carried out in the clinic for the duration another 6 weeks. The participants will be asked to keep diaries of their exercises they have carried out each week.
  Interventions: Other: core stability exercises

INTERVENTIONS:
Other: core stability exercises with teeth clenching — The intervention frequency will be 2 sessions per week for the duration of 6 weeks, comprising of 45 minutes session. Both groups will receive heat pack on lumbar spine for 12 minutes and both interventions will be held under the supervision of qualified Musculoskeletal Physiotherapists. During intervention and after 6 weeks of intervention.
  Arms: core stability exercises with teeth clenching
Other: core stability exercises — The intervention frequency will be 2 sessions per week for the duration of 6 weeks, comprising of 45 minutes session. Both groups will receive heat pack on lumbar spine for 12 minutes and both interventions will be held under the supervision of qualified Musculoskeletal Physiotherapists. During intervention and after 6 weeks of intervention.

SUMMARY:
Core stability strength & coordination is necessary to perform smooth & coordinated upper & lower extremity movements & function. Altered core stability muscle strength, coordination & poor motor control can cause low back pain (LBP). Physical therapists especially those working with children having neurodevelopmental problems or adults with neurological disorders such as stroke are aware of the concepts of global movements. In this concept, alterations in one body segment may bring changes in other body segments. In neurological rehabilitation, the concept of Neuro-Developmental Technique (NDT) introduced by Bobath got worldwide recognition. This concept states that there are specific key points in the neck, & shoulders that can facilitate normal movements by enhancing the activity of core musculature in functional movements for instance, sit to stand & walking. This concept was further explored by Burnstein and suggested that biomechanically body joints and motor control works together as functional unit and not as single limb movement. Bobath and proprioceptive neuromuscular facilitation (PNF) concepts further explained that movements of the eye, head and neck facilitate trunk movements. Electromyography studies have shown that both single and rhythmical jaw opening and closing movements not only produced well-coordinated jaw and head-neck movements but also produced atlanto-occipital and cervical spine joints movements. The author further concluded that mouth opening and closing in fetal yawning is associated with head extension-flexion movements indicating that functional connections between the jaw and head-neck is innate. A human jaw or masticatory system is connected to the motor system through cranial nerves unlike central motor system which is connected to the body through spinal motor system. Brainstem central pattern generator (CPG) control masticatory system through descending pathways and are involved in voluntary movements of the jaw such as mouth opening and closing. The higher brain centers cortical masticatory area and primary motor cortex control these movements. In the current back pain literature core stability exercises have been used in the management of chronic low back pain. The jaw is connected to the head-neck and neck is connected to the trunk. Therefore there is to study the effects of core stability exercises performed with and without jaw movements in the management of chronic low back pain.

DETAILED DESCRIPTION:
A randomized experimental controlled trial will be carried out to compare the effectiveness of core stabilization exercises performed with and without jaw movements in the management of nonspecific chronic low back pain. A total of 80 male and female volunteers having subjects with chronic nonspecific low back pain will be recruited in this study. All subjects will be assessed for transverse abdominal muscle strength contraction, pain and disability using Pressure Biofeedback Unit (BPU), Numeric Pain Rating Scale (NPRS 0-10cm) and Ronald Morris Disability Questionnaire (RMDQ 0-24) respectively. The scores on the mentioned scales will be documented as per guidelines. After baseline assessment, all subjects will be allocated to two groups through computer-generated random sampling. Group 1 will perform core stability exercises alone; Group 2 will perform core stability exercises with teeth clenching This study will be conducted at the Physiotherapy Department of Sindh Institute of Physical Medicine and Rehabilitation (SIPM&R). The computer-generated random sampling technique will be used to allocate the participants into the study groups. Data will be analyzed using SPSS 22 and one-way repeated measure ANOVA will be applied to see the mean difference in the 2 groups. For pair-wise comparison, the Tukey test will be applied. For pain and disability scales Friedman's test will be applied to see the two scales' median differences.

ELIGIBILITY:
Inclusion Criteria:

* · Participants having chronic low back pain lasting more than 12 weeks.

  * Age 20-45 years
  * Participants having nonspecific chronic low back pain with or without referred leg pain.
  * Both male and female patients.
  * Currently seeking care for low back pain.
  * No known TMJ pathology.
  * Had Magnetic Resonance Image (MRI) to exclude serious pathology and been diagnosed by the consultant and non-specific low back pain.

Exclusion Criteria:

* · Participants with known or suspected serious spinal pathology (fracture, metastatic, inflammatory or infective diseases of the spine, cauda equine syndrome/widespread neurological disorder, lumbar spondylosis, stenosis, spondylolisthesis).

  * Compromised nerve root
  * Previous spinal surgery or scheduled for major surgery during the treatment.
  * Co-morbid health conditions that would prevent active participation in the exercise programs such as asthma.
  * Low back pain having less than 12 weeks history.
  * Known Temporomandibular joint pathology or jaw pain.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | At baseline
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults, including those with chronic pain due to rheumatic diseases.
Numeric Pain Rating Scale | At 6th weeks
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults, including those with chronic pain due to rheumatic diseases.
Numeric Pain Rating Scale | At 12th weeks
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults, including those with chronic pain due to rheumatic diseases.
Roland Morris Questionnaire (RMQ): | At baseline
  RMQ is a standardized subjective assessment questionnaire that is used as Outcome tool to assess functional disability in acute and sub-acute low back pain.
Roland Morris Questionnaire (RMQ): | At 6th weeks
  RMQ is a standardized subjective assessment questionnaire that is used as Outcome tool to assess functional disability in acute and sub-acute low back pain.
Roland Morris Questionnaire (RMQ): | At 12th weeks
  RMQ is a standardized subjective assessment questionnaire that is used as Outcome tool to assess functional disability in acute and sub-acute low back pain.
Pressure Biofeedback unit (PBU): | At baseline
  Pressure Biofeedback unit (PBU) PBU is a reliable and valid tool for recording core stability muscle strength .
Pressure Biofeedback unit (PBU): | A 6th weeks
  Pressure Biofeedback unit (PBU) PBU is a reliable and valid tool for recording core stability muscle strength .
Pressure Biofeedback unit (PBU): | At 12th weeks
  Pressure Biofeedback unit (PBU) PBU is a reliable and valid tool for recording core stability muscle strength .

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Khan, MSAPT, Principal Investigator — University of Lahore
Locations (1):
- Sindh Institute of Physical Medicine & Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsao H, Druitt TR, Schollum TM, Hodges PW. Motor training of the lumbar paraspinal muscles induces immediate changes in motor coordination in patients with recurrent low back pain. J Pain. 2010 Nov;11(11):1120-8. doi: 10.1016/j.jpain.2010.02.004. PMID 20434958
- [Background] Sung PS. Disability and back muscle fatigability changes following two therapeutic exercise interventions in participants with recurrent low back pain. Med Sci Monit. 2013 Jan 14;19:40-8. doi: 10.12659/msm.883735. PMID 23314589
- [Background] Raine S, Meadows L, Lynch-Ellerington M. Bobath Concept: Theory and Clinical Practice in Neurological Rehabilitation. Wiley-Blackwell. 2009. 4- Bernstein, N. The Coordination and Regulation of Movement. Pergamon Press, Oxford. Bishop, B. 1967.
- [Background] Adler SS, Beckers D, Buck M. PNF in Practice: An Illustrated Guide. New York, NY: Springer. 2007.
- [Background] Voss DE, Ionta MK, Myers BJ. Proprioceptive Neuromuscular Facilitation. Patterns and Techniques. Philadelphia, PA: Harper & Row Publishers. 1985.
- [Background] HUMPHREY T. The spinal tract of the trigeminal nerve in human embryos between 7 1/2 and 8 1/2 weeks of menstrual age and its relation to early fetal behavior. J Comp Neurol. 1952 May;97(1):143-209. doi: 10.1002/cne.900970109. No abstract available. PMID 12981197
- [Background] Zafar H, Eriksson PO, Nordh E, Haggman-Henrikson B. Wireless optoelectronic recordings of mandibular and associated head-neck movements in man: a methodological study. J Oral Rehabil. 2000 Mar;27(3):227-38. doi: 10.1046/j.1365-2842.2000.00505.x. PMID 10784335
- [Background] Zafar H, Nordh E, Eriksson PO. Temporal coordination between mandibular and head-neck movements during jaw opening-closing tasks in man. Arch Oral Biol. 2000 Aug;45(8):675-82. doi: 10.1016/s0003-9969(00)00032-7. PMID 10869479
- [Background] Barry J. Sessle ,LimorAvivi-Arber, and Gregory M. Murray. Motor Control of Masticatory Muscles. Craniofacial Muscles: A New Framework for Understanding the Effector Side of Craniofacial Muscle Control. L.K. McLoon and F.H. Andrade (eds.) Toronto. 2013.
- [Derived] Khan M, Zafar H, Gilani SA, Farooqui WA, Ahmad A. The effects of lumbar stabilization exercises with and without jaw movements in non-specific low back pain (A randomized controlled trial). Pak J Med Sci. 2024 Jul;40(6):1116-1121. doi: 10.12669/pjms.40.6.9208. PMID 38952498